CLINICAL TRIAL: NCT03612596
Title: Narrative Visualization for Breast Cancer Survivors' Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17-0310; 1R21CA218543-01A1 (NIH)
Record Dates: First submitted 2018-07-25; First posted 2018-08-02 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: wearable; mobile app; physical activity; survivorship; narrative; identity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Narration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrative visualization (Experimental): Wearable activity monitor, app, and enhanced motivational scrapbook materials (instant camera, stickers, markers, enhanced content)
  Interventions: Behavioral: Narrative visualization
- Standard self-regulation (Active Comparator): Wearable activity monitor, app, and standard workbook materials (markers, a workbook with a calendar log to keep track of steps over time)
  Interventions: Behavioral: Standard self-regulation

INTERVENTIONS:
Behavioral: Narrative visualization — Participants use narrative visualization procedures to connect their step data to important events or feelings that occurred at the same time, then reflect on their behavior
  Arms: Narrative visualization
Behavioral: Standard self-regulation — Participants self-monitor steps using a wearable device, app, and a hand-written step log
  Arms: Standard self-regulation

SUMMARY:
This study tests the feasibility and acceptability of a physical activity intervention that combines use of a wearable activity monitor with a scrapbook. Half of the participants will receive this enhanced intervention, while the other half will receive a wearable activity monitor with a standard step log.

DETAILED DESCRIPTION:
Women breast cancer survivors could benefit from increased physical activity but are in need of greater motivation to be active. Interventions that use wearable activity monitors and mobile apps have shown promise in the short-term, but use drops off over time. Reports have suggested that users find the step data provided to be unclear and not very personally meaningful. The ultimate purpose of this line of research is to test whether enhanced motivational feedback, using scrapbooks, can increase motivation for activity. The scrapbooks will target integrated regulation, which is a type of motivation related to personal identity and values. Participants who receive this intervention will draw their step graph, add photographs and stickers an explanations to the graph, and answer reflection questions daily. Before testing the effects of this intervention on physical activity, the investigators must first ensure that the materials and procedures are feasible and acceptable. This small pilot study will allow the research team to iteratively test scrapbook materials and improve upon them for use in future studies. The investigators will compare an intervention using the enhanced materials to an intervention using only the wearable device, app, and a standard step log without scrapbook or reflection components. In addition to the primary outcome of feasibility (use of the scrapbook), the investigators will also explore the effects of the intervention on steps, motivational and values-related outcomes, and various aspects of feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 79 years
* Female
* Self-reported diagnosis of breast cancer
* BMI between 18 and 40 kg/m2
* Willingness to be randomized to any condition
* Participant is able to walk for exercise
* Able to read and understand English
* Daily access to a smartphone or similar device compatible with Garmin app
* PAR-Q+ indicates that physical activity would be safe (with note from physician required if any heart-related questions are endorsed)

Exclusion Criteria:

* Participant is active (150 minutes or more activity per week)
* Major health interventions (surgery, radiation, chemo) within the past 6 months
* Stroke, hip fracture, hip or knee replacement, or spinal surgery in the past 6 months
* History of orthopedic complications that would prevent optimal participation
* No active recurrence of cancer
* Self-reported smoker
* Reports psychological issues that would interfere with study completion (dementia, schizophrenia)
* Reports hospitalization within the past year due to psychiatric problem(s)
* Plans to be out of town for more than 2 weeks at a time during study period
* Clinical judgement concerning safety
* Currently participating in an organized commercial or research exercise program
* Another member of the household is a participant or staff member on this trial
* Current use of a wearable activity monitor

Ages: 55 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must self-report as women
Enrollment: 40 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Lyons, PhD, MPH, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide access to all data, regardless of publication, collected as a part of this project. All external investigators must submit a written request identifying their research question(s) and specifying the data they would like to analyze. The request must include a data security plan and explanation of how the data will be stored and who will have access. All requests will be reviewed by the investigators in conjunction with UTMB's Institute for Translational Sciences key resources (in particular, the regulatory and ethics resources) to be sure appropriate NIH requirements are followed.
Supporting Information: Study Protocol, SAP
Time Frame: Data will only be available upon request
Access Criteria: All external investigators must submit a written request identifying their research question(s) and specifying the data they would like to analyze. The request must include a data security plan and explanation of how the data will be stored and who will have access. All requests will be reviewed by the investigators in conjunction with UTMB's Institute for Translational Sciences key resources (in particular, the regulatory and ethics resources) to be sure appropriate NIH requirements are followed.

RESULTS

PARTICIPANT FLOW:
Period: 0 - 12 Weeks
Arm/Group | Narrative Visualization | Standard Self-regulation
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1
Period: 12 - 24 Weeks
Arm/Group | Narrative Visualization | Standard Self-regulation
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narrative Visualization | Standard Self-regulation | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (6.21) | 63 (4.86) | 62 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 16 | 19 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Daily Workbook Entries Completed
Description: Percentage of daily workbook entries completed out of the total possible number, measured by photography of intervention materials at 12 week assessment and then assessment of each page.
Time Frame: 12 weeks
Population: This outcome was only analyzed in the intervention group
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 20 | 0
percent | 44 (45) |

2. Secondary Outcome: Physical Activity as Measured by Steps Per Day During Intervention Period
Description: Mean of daily steps taken from accelerometers worn for 7 days
Time Frame: Change from 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 19 | 18
steps per day | 936.22 (1332.46) | 913.68 (1613.03)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.94, t-test, 2 sided

3. Secondary Outcome: Physical Activity as Measured by Daily Steps During No-intervention Maintenance Period
Description: Mean of steps per day taken from accelerometers worn for 7 days
Time Frame: Change from 12 to 24 weeks
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 19 | 18
steps per day | -829.37 (1320.50) | -893.73 (1191.96)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.88, t-test, 2 sided

4. Secondary Outcome: Intrinsic Regulation
Description: Self-reported intrinsic regulation on a scale from 0 (least motivated) to 4 (most motivated) using the Behavioral Regulation in Exercise Questionnaire - 3. Reported here are results from the intrinsic regulation subscale. Higher results on the scale indicate greater intrinsic regulation.
Time Frame: Change from 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 18 | 19
units on a scale | 0.49 (1.24) | 0.46 (1.03)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.94, t-test, 2 sided

5. Secondary Outcome: Integrated Regulation
Description: Self-reported integrated regulation on a scale from 0 (least motivated) to 4 (most motivated) using the Behavioral Regulation in Exercise Questionnaire - 3. Here, results from the integrated regulation subscale are reported. Higher numbers on the scale indicate greater integrated regulation.
Time Frame: Change from 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 18 | 19
units on a scale | 0.39 (1.13) | 0.17 (1.17)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.58, t-test, 2 sided

6. Secondary Outcome: Basic Psychological Needs: Autonomy
Description: Self-reported fulfillment of basic psychological needs on a scale from 1 (least fulfilled) to 5 (most fulfilled) using the Basic Psychological Needs in Exercise Questionnaire. The three subscales are perceived autonomy, competence, and relatedness. Here, autonomy is reported. A higher score means greater perceived autonomy.
Time Frame: Change from 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 18 | 19
units on a scale | 0.96 (1.17) | 0.50 (0.79)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.17, t-test, 2 sided

7. Secondary Outcome: Exercise Identity
Description: Self-reported identity as an exerciser on a scale from 1 (strongly disagree) to 7 (strongly agree) as measured by the Exercise Identity Scale. The two subscales are exercise beliefs and exercise role identity. Here, exercise role identity is reported. A higher score means greater exercise role identity.
Time Frame: Change from 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 18 | 19
units on a scale | 0.73 (1.42) | 0.48 (0.95)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.53, t-test, 2 sided; Please note that this analysis was not powered and was used to characterize effect size (d = 1.26) rather than test efficacy

8. Secondary Outcome: Basic Psychological Needs: Competence
Description: Self-reported fulfillment of basic psychological needs on a scale from 1 (least fulfilled) to 5 (most fulfilled) using the Basic Psychological Needs in Exercise Questionnaire. The three subscales are perceived autonomy, competence, and relatedness. Here, competence is reported. A higher score means greater perceived competence.
Time Frame: 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 19 | 18
units on a scale | 1.04 (1.25) | 0.77 (0.83)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.44, t-test, 2 sided; Please note that this analysis was not powered and was used to characterize effect size (d = 1.16) rather than test efficacy

9. Secondary Outcome: Basic Psychological Needs: Relatedness
Description: Self-reported fulfillment of basic psychological needs on a scale from 1 (least fulfilled) to 5 (most fulfilled) using the Basic Psychological Needs in Exercise Questionnaire. The three subscales are perceived autonomy, competence, and relatedness. Here, relatedness is reported. A higher score means greater perceived relatedness.
Time Frame: 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 19 | 18
units on a scale | 0.12 (1.36) | 0.41 (1.94)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.93, t-test, 2 sided; Please note that this analysis was not powered and was used to characterize effect size (d = 0.67) rather than test efficacy

10. Secondary Outcome: Self-reflection
Description: Self-reported self-reflection on a scale from 1 (strongly disagree) to 5 (strongly agree) using the Self-Reflection and Insight Scale. Here, we report changes in the insight subscale, which has 8 items and a range of 5-40. For this scale, higher values indicate greater levels of insight.
Time Frame: Change from 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 18 | 19
units on a scale | 0.56 (2.38) | 1.63 (3.58)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.29, t-test, 2 sided

11. Secondary Outcome: Quality of Life (Physical, Social, Emotional, Functional, and Breast Cancer-specific)
Description: Self-reported quality of life on a scale from 0 (not at all) to 4 (very much) using the Functional Assessment of Cancer Therapy - Breast measure. Reported here is the change in total score for the entire measure (with the total ranging from 0-123). Better quality of life is indicated by a lower score.
Time Frame: Change from 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 18 | 19
units on a scale | 4.04 (8.04) | 8.92 (12.13)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.16, t-test, 2 sided

12. Secondary Outcome: Importance of Valued Domains
Description: Self-reported importance of family, intimate relationships, friends, work, health, and growth values domains on a scale from 0 (not at all important) to 5 (extremely important) using the Chronic Pain Values Inventory. Reported here is the change in total across all domains, which is an average of the individual items (range: 0-5). A higher score indicates stronger endorsement of importance of the valued domains.
Time Frame: Change from 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 18 | 19
units on a scale | -0.23 (0.38) | 0.15 (0.56)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.02, t-test, 2 sided

13. Secondary Outcome: Success in Living According to Valued Domains
Description: Self-reported success in living according to values related to family, intimate relations, friends, work, health, and growth on a scale from 0 (not at all successful) to 5 (extremely successful) using the Chronic Pain Values Inventory. Reported here is the change in total across all domains, as an average across items (range: 0-5). A higher score indicates stronger endorsement of success in the valued domains.
Time Frame: Change from 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 18 | 19
units on a scale | 0.37 (0.74) | 0.48 (0.94)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.70, t-test, 2 sided

14. Secondary Outcome: Engaged Living
Description: Self-reported perception of living in accordance with one's values on a scale from 1 (completely disagree) to 5 (completely agree) using the Engaged Living Scale. The two subscales are valued living and life fulfillment. Reported here is the change in total results for the scale (which ranges from 16-80). Higher scores on this scale indicate higher levels of engaged living.
Time Frame: Change from 0 to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narrative Visualization | Standard Self-regulation
Number analyzed (Participants) | 18 | 19
units on a scale | 2.56 (6.64) | 3.39 (6.99)
Statistical Analysis 1: Comparison: Narrative Visualization vs Standard Self-regulation; Test type: Superiority; p = 0.71, t-test, 2 sided

15. Other Pre Specified Outcome: Receipt of Study Materials
Description: Self-reported percent of study materials received out of total supplied
Time Frame: 12 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Usefulness of Study Materials
Description: Self-reported usefulness of study materials, on a scale from 1 (strongly disagree they were useful) to 5 (strongly agree they were useful)
Time Frame: 12 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Participant Attrition
Description: Number of participants in each group who are lost to follow-up
Time Frame: 24 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Number of Serious Adverse Events
Description: The number of serious adverse events that occur during the intervention (0 - 12 weeks) and follow-up period (12 - 24 weeks)
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Days the Activity Monitor Was Worn
Description: The number of days the activity monitor was worn, as assessed via review of the mobile app
Time Frame: 12 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Completion of Values Clarification Activity
Description: From photographs taken of the intervention materials at the 12 week assessment, the investigators will assess whether participants in the enhanced intervention group completed their values clarification activity
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Narrative Visualization | Standard Self-regulation
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Missing data were imputed except for 3 participants with data missing at baseline. Results should be interpreted with caution due to the pilot nature of the trial and data collection occurring partially during spring/summer 2020.

Several outcomes (valued and engaged living, quality of life) were changed from secondary to other pre-specified, as these are likely not interpretable due to external factors (e.g., COVID-19 and social distancing).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT03612596/Prot_SAP_000.pdf